CLINICAL TRIAL: NCT07079163
Title: Comparison of Patient Satisfaction and Prosthetic Complications Between Conventional Immediate Surgical Obturators and 3D-printed Immediate Surgical Obturators With Enhanced Retention
Brief Title: Comparison of Conventional and 3D-printed Surgical Obturators for Maxillary Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma mahanna (Other)
Responsible Party: Sponsor-Investigator, Fatma mahanna, Assistant professor of prosthodontics, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A04011024RP
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Maxillary Defect Reconstruction
Keywords: Maxillary defects; Immediate surgical obturator; patient-centered outcomes; Digital; 3D-printed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Immediate Obturator Group/ obturator block (Experimental): Participants will receive a conventional immediate surgical obturator fabricated manually on a preoperative cast. Retention will be provided using clasps and/or wiring. The obturator will be inserted immediately after maxillectomy and used during the healing period.
  Interventions: Device: Obturator block
- Resin 3D-Printed Obturator Group (Experimental): Participants will receive a resin 3D-printed immediate surgical obturator, digitally designed using intraoral scans and CBCT data. Retention will be achieved using 3D-printed clasps and palatal screws. The obturator will be inserted immediately after surgery and monitored during healing.
  Interventions: Device: Obturator block
- Metallic 3D-Printed Obturator Group (Experimental): Participants will receive a metallic 3D-printed immediate surgical obturator, digitally designed using fused CBCT and digital impressions. The prosthesis will include metal clasps and palatal screws for enhanced retention. It will be delivered at surgery and assessed over the healing period.
  Interventions: Device: Obturator block

INTERVENTIONS:
Device: Obturator block — A manually fabricated obturator using a preoperative maxillary cast, retained with clasps and wire. Delivered immediately after maxillectomy.
  Other Names: Conventional Immediate Obturator Group
  Arms: Conventional Immediate Obturator Group/ obturator block
Device: Obturator block — A digitally designed obturator based on fused CBCT and intraoral scan data. Fabricated in resin using 3D-printing, and retained with 3D-printed clasps and palatal screws. Delivered immediately post-maxillectomy
  Other Names: Resin 3D-Printed Surgical Obturator
  Arms: Resin 3D-Printed Obturator Group
Device: Obturator block — A digitally designed and 3D-printed obturator fabricated in metal, using CBCT and intraoral scan data. Retention is provided by metal clasps and palatal screws. Delivered during or immediately after surgery.
  Other Names: Metallic 3D-Printed Surgical Obturator
  Arms: Metallic 3D-Printed Obturator Group

SUMMARY:
This randomized controlled clinical trial aims to compare patient satisfaction and prosthetic complications associated with three types of immediate surgical obturators used in maxillectomy patients. A total of 24 patients with acquired maxillary defects will be randomly assigned to receive one of three obturator designs: (1) conventional obturators retained with clasps and wire, (2) resin 3D-printed obturators with printed clasps and palatal screws, or (3) metallic 3D-printed obturators with metal clasps and palatal screws.

Patient satisfaction will be evaluated using the Obturator Functioning Scale (OFS), and postoperative complications such as discomfort, lack of retention, or mucosal irritation . The study seeks to determine whether digital fabrication and enhanced retention methods improve clinical outcomes compared to traditional approaches

DETAILED DESCRIPTION:
Maxillary defects resulting from maxillectomy procedures lead to significant impairments in speech, mastication, swallowing, and quality of life. Rehabilitation typically involves either surgical reconstruction or the use of a prosthetic obturator. Immediate surgical obturators (ISOs) are commonly used during or immediately after surgery to seal the oronasal communication and support healing. However, conventional obturators are often bulky, manually fabricated, and prone to poor retention due to tissue changes during early healing, leading to reduced patient satisfaction and increased complications.

Recent advancements in digital technology, including intraoral scanning and cone beam computed tomography (CBCT), allow for the precise design and 3D printing of obturators customized to the anticipated defect. Enhanced retention strategies such as palatal screws and custom clasps may offer improved stability, function, and comfort compared to conventional designs.

This randomized controlled clinical trial aims to evaluate and compare the clinical performance of three types of immediate surgical obturators in patients undergoing maxillectomy. A total of 24 patients with acquired maxillary defects and sufficient remaining dentition will be randomly assigned to one of three groups:

Group I: Conventional obturators retained with clasps and wire

Group II: Resin 3D-printed obturators with printed clasps and palatal screws

Group III: Metallic 3D-printed obturators with metal clasps and palatal screws

The study's primary outcome is patient satisfaction, assessed using the Obturator Functioning Scale (OFS), which evaluates prosthesis-related comfort, appearance, speech, and function. Secondary outcomes include postoperative prosthetic complications such as pain, ulceration, poor fit, or dislodgement. Assessments will be conducted during the standard healing period.

This study will provide valuable insights into the impact of digital workflows and retention techniques on the functional performance and patient-centered outcomes of obturator prostheses following maxillectomy. Ethical approval has been obtained, and all participants will provide informed consent prior to inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for maxillectomy with the remaining number of teeth
* Referral to Maxillofacial Prosthodontic Unit, Mansoura University

Exclusion Criteria:

* contraindication to surgery (not physically fit to underwent surgery)

Ages: 36 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 2-3 weeks after surgery
  Patient satisfaction: measured by Obturator Functioning Scale (OFS) over 2-3 weeks.The Obturator Functioning Scale (OFS) is a patient-reported outcome measure developed to assess the functional performance and satisfaction with an obturator prosthesis, particularly in maxillectomy patients. It evaluates multiple domains related to oral rehabilitation.The OFS typically includes items addressing the following:
  Appearance (Esthetics)
  Speech Intelligibility
  Swallowing (Deglutition)
  Chewing/Mastication
  Comfort
  Retention and Stability
  Overall Satisfaction 5-point Likert scale (e.g., 1 = very poor, 5 = excellent

SECONDARY OUTCOMES:
complications | 2-3 weeks after surgery
  Postoperative complications: type and frequency (pain, discomfort, dislodgement, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: fatma mahanna, Phd, Study Chair — Mansoura university, faculty of dentistry
Locations (1):
- Maxillofacial Prosthodontic Unit, Faculty of Dentistry, Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided